CLINICAL TRIAL: NCT02771353
Title: The HeartSpare Plus 1B Trial: A Randomised Phase II Trial Comparing the Resource Impact, Acute Toxicity and Feasibility of Different Pan-lymph Node Radiotherapy Techniques for Breast Cancer Patients
Brief Title: The HeartSpare Plus 1B Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCR4501
Record Dates: First submitted 2016-04-26; First posted 2016-05-13 (Estimated); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- WT_vDIBH (Active Comparator): Wide tangent radiotherapy in voluntary deep inspiratory breath hold
  Interventions: Radiation: WT_vDIBH
- VMAT_FB (Active Comparator): Volumetric modulated arc therapy in free breathing.
  Interventions: Radiation: VMAT_FB

INTERVENTIONS:
Radiation: WT_vDIBH
  Arms: WT_vDIBH
Radiation: VMAT_FB
  Arms: VMAT_FB

SUMMARY:
This study aims to compare the resource impact, acute toxicity and feasibility of different pan-lymph node radiotherapy techniques. Radiotherapy using wide tangents with the patient in breath hold will be compared against volumetric modulated arc therapy (VMAT) in free breathing in the main trial. A parallel study will asses the accuracy of VMAT treatments using voluntary deep inspiratory breath hold compared to an active breathing controlled breath hold device.

DETAILED DESCRIPTION:
Following publication of results of two large randomised clinical trials, pan-lymph node radiotherapy (pan-LN RT) (including treatment of the internal mammary chain) is set to become standard treatment in patients with lymph-node positive breast cancer. Traditional pan-LN RT techniques deliver high radiation doses to the heart and lungs which can cause long-term side-effects in women many years after their treatment. Modern techniques including breath-holding and volumetric-modulated arc therapy (VMAT) can reduce doses to heart and lungs but the investigators do not yet know which technique(s) are best in terms of resource costs, short to medium-term side-effects, and day to day accuracy. This study will compare the time taken to deliver pan-LN RT using breath-holding versus VMAT and will collect side-effect data up to one year following treatment as well as modelling long-term cardiac risks based on heart doses delivered. The results of the main study will help guide clinicians and departments in selecting the best pan-LN RT techniques for their patients. A parallel study will evaluate the combination of breath-hold and VMAT using a machine-based technique called the active-breathing controlled (ABC) device against a more simple voluntary breath-hold technique were patients simply take a breath in and hold it for up to 20 seconds at a time. These techniques will be compared in terms of their day-to-day accuracy. If the simpler technique proves as accurate as the ABC-technique, this will establish the simpler technique as a less resource-intensive standard of care adoptable by other radiotherapy departments.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Female or male
* Invasive carcinoma of the breast (left or right-sided)
* Breast conservation surgery or mastectomy
* Axillary staging and/or dissection
* pT1-T4,N1-2,M0 disease
* Histological involvement of axillary lymph nodes
* Indication for radiotherapy to the IMC, axillary levels I-III and/or level IV
* Patient able to tolerate breath hold
* Performance status 0-1

Exclusion Criteria:

* Contralateral and/or previous ipsilateral breast cancer, irrespective of date of diagnosis
* Past medical history of malignancy except (i) basal cell skin carcinoma, (ii) CIN cervix uteri, (iii) non-breast malignancy allowed if treated with curative intent and at least 5 years disease free
* Previous radiotherapy to any region above the diaphragm

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2016-12-12 (Actual); Primary Completion 2019-01-15 (Actual); Study Completion 2019-01-15 (Actual)

PRIMARY OUTCOMES:
Linear Accelerator time | 3 weeks
  Patient mounting couch to linear accelerator being turned off

SECONDARY OUTCOMES:
Acute toxicity - Skin | 5 weeks
  CTCAE grading
Acute toxicity - lung (pneumonitis) | 5 weeks
  CTCAE grading
Acute toxicity - oesophagitis | 5 weeks
  CTCAE grading
Acute toxicity - fatigue | 5 weeks
  EORTC QLQ-C30 + FA13
Acute toxicity - quality of life | 5 weeks
  EORTC QLQ-C30 + BR23
Intermediate toxicity - lung (pneumonitis) | up to 1 year
  CTCAE pneumonitis assesment
Intermediate toxicity - fatigue | up to 1 year
  EORTC QLQ-C30 + FA13
Intermediate toxicity - quality of life | up to 1 year
  EORTC QLQ-C30
Intermediate toxicity - lymphoedema/ shoulder dysfunction | up to 1 year
  EORTC BR23
Organ at risk dose - ipsilateral lung | Immediate
  mean dose to the ipsilateral lung (Gy) measured using DVH
Organ at risk dose - contralateral lung | Immediate
  mean dose to the contralateral lung (Gy) measured using DVH
Organ at risk dose - heart | Immediate
  mean dose to the heart (Gy) measured using DVH
Organ at risk dose - contralateral breast | Immediate
  mean dose to the contralateral breast (Gy) measured using DVH
Organ at risk dose - thyroid | Immediate
  mean dose to the thyroid (Gy) measured using DVH
Organ at risk dose - humeral head | Immediate
  mean dose to the humeral head (Gy) measured using DVH
Organ at risk dose - brachial plexus | Immediate
  maximum dose to the brachial plexus (Gy) measured using DVH
Organ at risk dose - Left anterior descending coronary artery | Immediate
  maximum dose to the Left anterior descending coronary artery (Gy) measured using DVH
Organ at risk dose - oesophagus | Immediate
  maximum dose to the oesophagus (Gy) measured using DVH
Time taken to plan and check radiotherapy | Immediate
Inter-fraction reproducibility | 3 weeks
  Distance - shift from planning CT on CBCT (mm)

IPD SHARING:
Plan to Share IPD: Yes